CLINICAL TRIAL: NCT06978946
Title: Clinical Efficacy and Safety of Deep Cervical Lymphaticovenous Anastomosis (DLVA) in Moderate-to-Severe Neurodegenerative Dementia
Brief Title: Deep Cervical Lymphaticovenous Anastomosis Surgery for Moderate-to-Advanced Dementia Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wang Gang, Professor, RenJi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLVA-NDD-01
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Lewy Body Dementia (LBD); Frontotemporal Dementia (FTD); Dementia; Parkinsons Disease With Dementia (PDD)
Keywords: Alzheimer Diseas; Lewy Body Dementia (LBD); Frontotemporal Dementia (FTD); Lymphaticovenous Anastomosis; Parkinsons Disease
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia; Dementia; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (No Intervention): This group served as the control group, consisting of AD patients who received no intervention.
- PDD surgical intervention group (Experimental): Participants in this group will undergo the Deep Cervical Lymphaticovenous Anastomosis (DLVA) surgery.
  Interventions: Procedure: Deep Cervical Lymphaticovenous Anastomosis(DLVA)
- DLB surgical intervention group (Experimental): Participants in this group will undergo the Deep Cervical Lymphaticovenous Anastomosis (DLVA) surgery.
  Interventions: Procedure: Deep Cervical Lymphaticovenous Anastomosis(DLVA)
- FTD surgical intervention group (Experimental): Participants in this group will undergo the Deep Cervical Lymphaticovenous Anastomosis (DLVA) surgery.
  Interventions: Procedure: Deep Cervical Lymphaticovenous Anastomosis(DLVA)
- AD surgical intervention group (Experimental): Participants in this group will undergo the Deep Cervical Lymphaticovenous Anastomosis (DLVA) surgery.
  Interventions: Procedure: Deep Cervical Lymphaticovenous Anastomosis(DLVA)

INTERVENTIONS:
Procedure: Deep Cervical Lymphaticovenous Anastomosis(DLVA) — This surgery will enhance the drainage of cerebral lymphatic fluid by surgically establishing a connection between lymphatic vessels and veins in the neck
  Arms: AD surgical intervention group; DLB surgical intervention group; FTD surgical intervention group; PDD surgical intervention group

SUMMARY:
This clinical trial aims to evaluate the clinical efficacy and safety of Deep Cervical Lymphaticovenous Anastomosis (DLVA) in patients aged 50-80 with moderate to severe neurodegenerative dementia. Participants will undergo surgical treatment, followed by cognitive assessments, PET/MRI scans, lymph fluid/cerebrospinal fluid collection, and blood tests. Additionally, the study will perform an in-depth analysis of DLVA's therapeutic mechanisms using multimodal imaging and molecular biology experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50-80 years
2. AD participants meet the diagnostic criteria for Alzheimer's disease established by the National Institute on Aging and the Alzheimer's Association (NIA-AA); FTD participants meet the diagnostic criteria defined by the International Consortium on FTD; DLB participants meet the 2017 diagnostic criteria of the DLB Consortium; PDD participants meet the 2007 diagnostic criteria of the Movement Disorder Society or the 2011 Chinese diagnostic guidelines for PDD;
3. Mini-Mental State Examination (MMSE)<than 21, Montreal Cognitive Assessment (MoCA) score<17, and Clinical Dementia Rating (CDR) score ≥2;
4. Diagnosed by clinicians as having moderate to severe disease;
5. On stable medication regimen for ≥1 month
6. Signed informed consent and demonstrated good compliance

Exclusion Criteria:

1. Dementia caused by other conditions, including: vascular dementia; central nervous system infections due to HIV, syphilis, etc.; Creutzfeldt-Jakob disease; Huntington's disease; traumatic brain injury-related dementia; dementia due to toxic or alcohol-related factors; major systemic diseases such as hepatic or pulmonary encephalopathy; subdural hematoma; endocrine disorders such as thyroid or parathyroid disease; vitamin deficiency; or any other cause of dementia.
2. Presence of severe or unstable medical conditions, including but not limited to cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, neurological (excluding cognitive impairment), psychiatric, immunological, or hematological disorders, or any other condition deemed by the investigator to potentially interfere with study results; or life expectancy < 24 months.
3. Current diagnosis of any primary psychiatric disorder other than cognitive impairment. If, in the investigator's opinion, the psychiatric condition or symptoms may interfere with cognitive assessment or the subject's ability to complete the study, exclusion is required. Subjects with a history of schizophrenia or other chronic psychotic disorders should also be excluded.
4. Contraindications to deep cervical LVA surgery, including left vagus nerve injury, severe infection at the surgical site, significant dysfunction of the heart, lungs, liver, kidneys, or other organ systems, a history of head and neck radiation therapy or surgery, preoperative anesthetic evaluation of ASA grade III or above, or inability to tolerate prolonged surgery.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Severity of dementia | preoperative day 3，postoperative day 3、month 3、month 6、month12
  Measured using the (Clinical Dementia Rating Scale - Sum of Boxes(CDR-SB).The CDR-SB is a quantitative tool used to assess the severity of cognitive and functional impairment across six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a scale from 0 (no impairment) to 3 (severe impairment), resulting in a total CDR-SB score ranging from 0 to 18. A score of 0 indicates no dementia, scores between 0.5 and 4.0 suggest very mild cognitive impairment or mild cognitive decline, 4.5 to 9.0 corresponds to mild dementia, 9.5 to 15.5 reflects moderate dementia, and scores between 16 and 18 represent severe dementia. In general, higher CDR-SB scores reflect greater cognitive and functional impairment, while lower scores indicate better cognitive performance and daily functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No